CLINICAL TRIAL: NCT06234332
Title: Peking University Birth Cohort in Weifang
Brief Title: Peking University Birth Cohort in Weifang (PKUBC-WF)
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Hai-Jun Wang, Prof., Peking University
Other Study IDs: PKUBC-WF
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Health Problems in Pregnancy; Pregnancy Outcomes; Gestational Diabetes; Gestational Hypertension; Preterm Birth; Obesity; Mother-Infant Interaction; Child Development; Anemia
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced; Premature Birth; Obesity; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pregnancy:
  During pregnancy and 42 days after delivery: the remaining peripheral blood sample (about 2ml) and urine sample (about 8ml); additional anticoagulant peripheral blood (5ml) and urine (10ml) of women and their husband (only when pregnant women were enrolled) .
  Pre-delivery: feces (5g).
  After delivery: samples of umbilical cord blood (about 10ml), placenta (8 to 10 pieces of tissue with a diameter of 1.0cm), umbilical cord (4 pieces of tissue with a length of 1cm), meconium (5g), and heel blood (about 0.5ml)
  Childhood:
  6 months of age: extra fingertip blood (about 0.5ml). At the age of 1 and 2: urine sample (about 10ml) . At the age of 3 and 6: the remaining peripheral blood sample (about 2ml) and urine sample (about 8ml) .
  At the age of 9, 12, 15 and 17: the remaining peripheral blood sample examined by blood biochemistry (about 2ml) , the remaining peripheral blood sample examined by blood routine (about 2ml) and urine routine residual urine sample (about 8ml).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure group: Group with environmental, nutritional or lifestyle exposures
  Interventions: Other: No Interventions
- Non-exposed group: Group without any environmental, nutritional and lifestyle exposures

INTERVENTIONS:
Other: No Interventions — No intervention This is an observational study without any intervention
  Groups: Exposure group

SUMMARY:
The PKUBC-WF is a prospective cohort study carried out in Weifang city of Shandong, China. The primary aim of this study is to investigate the short-term and long-term effects of pre-pregnant and prenatal exposure on maternal and child health. Data are collected regarding environmental, nutritional and lifestyle exposures as well as short-term and long-term health outcomes of mothers and their children from birth to before 18 years old. Biological samples including peripheral blood, urine, placenta, umbilical cord, cord blood, and faeces are also collected.

DETAILED DESCRIPTION:
Maternal and child health is of great concern globally. Early life phase of a fetus and infant is a critical period for the development of health and disease in the whole life. Exposure of negative environmental, nutritional and lifestyle factors in pregnant women during this period can have adverse effects on fetal and infant. In addition, for mothers, complications during pregnancy could also have a negative effect on long-term health of mothers, such as diabetes, hypertension. Thus, the Peking University Birth Cohort in Weifang is primarily aimed to investigate the short-term and long-term effects of pre-pregnant and prenatal exposure on maternal and child health. Data are collected regarding environmental, nutritional and lifestyle exposures as well as short-term and long-term health outcomes of mothers, husbands and their children from birth to before 18 years old. Biological samples including peripheral blood, urine, placenta, umbilical cord, cord blood, and faeces samples are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman

  1. Pregnant women, 6-13^+6 gestational weeks
  2. Resided in Weifang in the past half years and have no plan to move out after delivery
  3. Pregnant women who plan to have antenatal care and delivery in Weifang maternal&Child Hospital.
  4. Pregnant women who is willing to participate in this study with informed consent
* Pregnant woman's husband

  1. His wife was eligible for enrollment
  2. He is the biological father of the child (his wife's current pregnancy)
  3. Pregnant women's husband who is willing to participate in this study with informed consent
* Offspring 4. Children born to pregnant women who met the inclusion criteria after enrolling in this study.

  5. Before the age of 8 years, his/her mother provided written informed consent. 6. After 8 years old, he/she agreed to continue this study and signed the informed consent.

Exclusion Criteria:

* Participants who cannot communicate normally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women and their children in Weifang, China
Sampling Method: Non-Probability Sample
Enrollment: 2800 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Numbers and morbidity of participants with pregnancy complications | At delivery
  Including gestational diabetes, gestational hypertension, anemia, and hypothyroidism during pregnancy
Numbers and morbidity of participants with adverse pregnancy outcomes | At delivery
  Including preterm birth, low birth weight, macrosomia, abortion, stillbirth, and birth defects.

SECONDARY OUTCOMES:
Weight in kilogram changes during childhood | At birth and age at 6 weeks, 6 months, 12 months, 2 years, 3 years, 6 years, 9 years, 12 years, 15 years, and 17 years
  Measured by health professionals in clinic
Height in centimeter changes during childhood | At birth and age at 6 weeks, 6 months, 12 months, 2 years, 3 years, 6 years, 9 years, 12 years, 15 years, and 17 years
  Measured by health professionals in clinic
Early Child development | Age at 6 weeks, 6 months and 12 months
  Measured by Ages&Stages Questionnaires (ASQ).There are 6 questions in each of 5 domains of development: communication, gross motor, fine motor, problem-solving skills, and adaptive skills. Each question is given a 10 (yes), 5 (sometimes), or 0 (not yet) score according to the parents' answers. The sum scores (range from 0 to 300) and scores for each domain (range from 0 to 60) are calculated. Chinese norms are available for each domain, and any domain screened <2 SDs below the mean is considered a positive screening. A higher ASQ score means better development.
Incidence of diabetes mellitus in women | 6 weeks after delivery and 3 years after delivery
  Measured by health professionals in clinic
Incidence of hypertension in women | 6 weeks after delivery and 3 years after delivery
  Measured by health professionals in clinic
Incidence of child overweight and obesity | At birth and age at 6 weeks, 6 months, 12 months, 2 years, 3 years, 6 years, 9 years, 12 years, 15 years, and 17 years
  Measured by health professionals in clinic
Incidence of autism spectrum disorder in children | Age at 2 years, 3 years
  Measured by The Modified Checklist for Autism in Toddlers, Revised with Follow-Up (M-CHAT-R/F) and Autism Behavior Checklist (ABC) scales
Incidence of attention-deficit/hyperactivity disorder in children | Age at 6 years
  Measured by The Child Behavior Checklist (CBC) scale
Incidence of anxiety in adolescents | Age at 9 years, 12 years, 15 years, and 17 years
  Measured by Social Anxiety Scale for Adolescents (SAS-A) scale
Incidence of depression in adolescents | Age at 9 years, 12 years, 15 years, and 17 years
  Measured by Beck Depression Inventory-II (BDI-II) scale

CONTACTS AND LOCATIONS:
Overall Officials: Haijun Wang, Ph.D, Principal Investigator — Peking University
Locations (1):
- Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No